CLINICAL TRIAL: NCT01497821
Title: A Phase 1 First-in-Human Study Evaluating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 172 in Subjects With Relapsed / Refractory Renal Cell Carcinoma
Brief Title: AMG 172 First in Human Study in Patients With Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20090515
Record Dates: First submitted 2011-12-16; First posted 2011-12-23 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Renal Cell Adenocarcinoma; Clear Cell Renal Carcinoma; Clear Cell Renal Cell Carcinoma; Renal Cell Carcinoma
Keywords: Amgen; Phase 1; First in Human; Relapsed / Refractory Renal Cell Carcinoma (RCC); Kidney Cancer; Clinical Trial; Antibody drug conjugate (ADC); Open-label; Oncology
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasms

ARMS (2):
- Dose exploration (Experimental): Pre-specified nominal doses are proposed in the dose exploration at two dosing frequencies: every two weeks and every three weeks. Intermediate doses may also be used if required based on the Continuous Reassessment Method (CRM) design.
  Interventions: Drug: AMG 172
- Dose expansion (Experimental): Dose and dosing frequency selected from Part 1 dose exploration.
  Interventions: Drug: AMG 172

INTERVENTIONS:
Drug: AMG 172 — AMG 172 is an antibody drug conjugate

SUMMARY:
This is the first-in-human (Phase I) study of AMG 172, an antibody drug conjugate (ADC), in subjects with kidney cancer [Clear Cell Renal Cell Carcinoma (ccRCC)] who have relapsed or who have refractory disease following at least two prior therapies. The purpose of the study is to evaluate safety and pharmacokinetics (PK) of AMG 172, and also evaluate the objective response rate in patients with ccRCC receiving AMG 172. The study will be conducted in two Parts: Part 1 will explore doses of AMG 172 given every two weeks and every three weeks to determine the safety, tolerability and pharmacokinetics to establish a maximum tolerated dose (MTD), and Part 2 (dose expansion) will examine safety, tolerability, PK and overall response rate in subjects treated at the MTD established in Part 1 for either every two week or every three week dosing.

DETAILED DESCRIPTION:
This First in- human study of AMG 172 will be conducted in two parts: Part 1 (dose exploration) and Part 2 (dose expansion). Part 1 of the study is aimed at evaluating the safety, tolerability and PK of AMG 172 given every two weeks and every three weeks in subjects with relapsed / refractory cc RCC, and Part 2 is aimed at evaluating safety, tolerability, PK and response rate in subjects treated at the MTD established in Part 1 for either every two week or every three week dosing. Up to 48 subjects may be enrolled in Part 1, and up to 30 subjects may be enrolled in Part 2. The dose of AMG 172 utilized in Part 2 will be dependent upon data obtained in Part 1 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a pathologically documented, definitively diagnosed, clear cell RCC that is relapsed/refractory following at least two lines of systemic therapy (one of which must be a tyrosine kinase), or the subject refuses standard therapy
* Measurable disease per RECIST 1.1 criteria. Subjects with non-measurable, but evaluable disease are also eligible for Part 1 of the study.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1
* Willing to provide tumor samples and / or slides
* Hematological function, as follows:

  1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L;
  2. Platelet count ≥ 100 x 10^9/L;
  3. Hemoglobin > 9 g/dL
* Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 x institutional upper limit of normal (IULN)
* Hepatic function, as follows:

  1. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x ULN;
  2. Total bilirubin < 1.5 x ULN (< 3.0 x ULN for subjects with documented Gilbert's Disease or for whom the indirect bilirubin level suggests an extrahepatic source of elevation);
  3. Alkaline phosphatase < 2 x ULN (< 5 x ULN in subjects whom the PI and sponsor agree that clinical data suggest extrahepatic source of elevation)
* Other inclusion criteria may apply

Exclusion Criteria:

* Known primary central nervous system (CNS) tumors or brain metastases
* History of bleeding diathesis
* Myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication, or uncontrolled hypertension in the opinion of the investigator
* Clinically significant ECG changes which obscure the ability to assess the PR, QT, and QRS interval; congenital long QT syndrome
* A baseline ECG QTcF > 470 msec
* Known positive test for human immunodeficiency virus (HIV)
* Known acute or chronic hepatitis B or hepatitis C infection as determined by serologic tests
* Other exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Clinically significant or ≥ Grade 3 CTCAE changes in safety laboratory tests, physical examinations, ECGs, or vital signs | 28 days after the last subject enrolled of each cohort in Part 1 and every 10 subjects enrolled in Part 2 (if available)
PK parameters including but not limited to, maximum observed concentration (Cmax), area under the concentration-time curve (AUC) and half life (t1/2) | 12 time points up to 8 weeks
Objective response rate for subjects treated at MTD based on RECIST 1.1 | 3 years
The MTD for at least one of two dosing schedules: every two weeks or every three weeks | 3 years

SECONDARY OUTCOMES:
Development of human anti-human antibody against AMG 172 | 1 year
Objective response rate for subjects not treated at MTD based on RECIST 1.1 | 3 years
Clinical benefit as measured by duration of response per RECIST 1.1 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (2):
  - Research Site, Scottsdale, Arizona
  - Research Site, St Louis, Missouri
- Research Site, Villejuif, France
- Research Site, Heidelberg, Germany

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com